CLINICAL TRIAL: NCT02861625
Title: CONDOL01: Evaluation on the Experience of Bereavement, of a Medical Consultation, Proposed by a Letter of CONDOLence to the Patients' Relatives Versus Standard Practice After the Death of the Patient: A Multicenter, Randomized Trial
Brief Title: CONDOL01: Evaluation on the Experience of Bereavement, of a Medical Consultation, Proposed by a Letter of CONDOLence to the Patients' Relatives Versus Standard Practice After the Death of the Patient
Acronym: CONDOL01
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: CONDOL01-IPC 2015-006
Record Dates: First submitted 2016-08-01; First posted 2016-08-10 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Caregivers

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: letter of condolence offering to the reliable person a post-death consultation with the reference physician (sent between J15 and J30 post death)
  Interventions: Behavioral: Letter of condolence and post-death medical consultation
- Group B: no intervention, i.e without a letter of condolence proposing a consultation with the reference physician

INTERVENTIONS:
Behavioral: Letter of condolence and post-death medical consultation — Process of sending a letter of condolence with consultation proposition.
  Groups: Group A

SUMMARY:
The aim of this randomized multicenter study is to evaluate the impact in offering the condolence letter to the family caregivers (indicated as the reliable person by the patient himself at each hospitalization) and a bereavement consultation with the reference physician.

DETAILED DESCRIPTION:
The hypothesis is that offering the opportunity to clarify questions about the patients' terminal care will influence positively the grieving process. In particular, the study team hypothesized that psychological morbidity will be reduced (main objective) as well as some aspects of QOL (secondary objective). It is also assumed that the situations of conflict (solicitations for medical records, number of legal procedures) will be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Patient died in the institution
* Patient for which the reliable person has been identified
* Acceptation of the reference physician to send a letter of condolence with the proposed consultation

Exclusion Criteria:

* The physician already met with the caregiver after the patient's death

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of the reliable person (a family member and/or caregiver, designed by the patient himself at each hospitalization) of cancer patients who have died in one of the participating center.
Sampling Method: Probability Sample
Enrollment: 432 (Estimated)
Dates: Start 2018-05-24 (Actual); Primary Completion 2022-06-04 (Estimated); Study Completion 2022-06-04 (Estimated)

PRIMARY OUTCOMES:
Evolution of mental component score (MCS) of the SF-36 questionnaire | 3 months post death
  It will be evaluated by self-questionnaires send at 3 months after the death of the patient, in the 2 groups (with or without condolence letter proposing a post-death consultation).

SECONDARY OUTCOMES:
Quality of life of the caregivers after the death of the patient evaluated by specific caregivers CarGOQoL questionnaire | 1 year post death
Quality of life of the caregivers after the death of the patient evaluated by SF36 questionnaire | 1 year post death
Anxiety of the caregivers after the death of the patient | 1 year post death
  Evaluated by Spielberger State Trait anxiety questionnaire
Depression of the caregivers after the death of the patient | 1 year post death
  Evaluated by Hospital Anxiety and Depression Scale
Complicated grief | 1 year post death
  Evaluated by Inventory of complicated grief questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gwenaelle Gravis, MS, Principal Investigator — Institut Paoli-Calmettes
Locations (2):
- France (2):
  - Institut Paoli Calmettes, Marseille, Bouches Du Rhone
  - GRAVIS, Marseille